CLINICAL TRIAL: NCT06424106
Title: Effect of Glucagon on Fasting Insulin Secretion and Glucose Metabolism in Subjects Without Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 24-002639
Record Dates: First submitted 2024-05-13; First posted 2024-05-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: PreDiabetes
Keywords: Insulin secretion; glucagon secretion; endogenous glucose production; glucose disappearance
MeSH Terms: conditions — Prediabetic State | interventions — Glucagon; Glucose

STUDY DESIGN:
Intervention Model Description: All participants will complete two experiments conducted in random order. On one day they will receive a graded glucagon infusion while on the other they will receive a glucose infusion that replicates the glucose concentrations observed in the first study day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucagon Infusion (Active Comparator): A glucagon infusion (0.2 ng/kg/min) will start at 0900 (0 min), increasing to 0.4 (1000), 0.6 (1100) and 0.8 ng/kg/min (1200) at 60-minute intervals - ending at 1300 (240 min).
  Interventions: Other: Glucagon
- Glucose Infusion (Placebo Comparator): At 0900 (0 min) a glucose infusion will commence, and the infusion rate varied to replicate (± 5mg/dL) that individual's glucose concentrations observed during the Glucagon Infusion Day. The experiment will end at 1300 (240 min) when infusions are stopped.
  Interventions: Other: Glucose

INTERVENTIONS:
Other: Glucagon — a variable rate glucagon infusion
  Arms: Glucagon Infusion
Other: Glucose — a variable rate glucose infusion
  Arms: Glucose Infusion

SUMMARY:
Fasting hyperglycemia contributes disproportionately to nonenzymatic glycosylation and the microvascular complications of type 2 diabetes. However, little is known about the regulation of glucose concentrations in the fasting state relative to what is known about the postprandial state. The proposed experiment is part of a series of experiments designed to establish how glucagon and insulin interact with their receptors to control fasting glucose in health and in prediabetes.

DETAILED DESCRIPTION:
The interaction between α-cell and β-cell function to regulate fasting glucose is incompletely understood. This is an important gap in our knowledge as fasting glucose contributes disproportionately to HbA1c and the microvascular complications of type 2 diabetes (T2DM). The regulation of fasting glucose in health and disease is relatively understudied.

Insulin and glucagon should regulate glucose reciprocally through direct interaction; insulin restrains α-cell secretion while glucagon directly stimulates β-cell secretion. In addition, there are indirect interactions via changes in glucose. Glucagon increases endogenous glucose production (EGP) increasing glucose (and insulin secretion). Conversely, insulin stimulates glucose disappearance (Rd) and suppresses EGP, lowering glucose (and stimulating glucagon).

However, this does not appear to occur uniformly in prediabetes. For example, in impaired fasting glucose (IFG), glucagon secretion rate (GSR) is inappropriate for the prevailing glucose. This is not accompanied by reciprocal changes in insulin secretion rate (ISR). Variability in the hepatic response to glucagon and to insulin further compound the dysregulation of fasting glucose. The net effect of these variables is unknown. This experiment is intended to test the hypothesis that impaired glucagon-induced insulin secretion contributes to fasting hyperglycemia in IFG.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with normal or impaired fasting glucose and normal or impaired glucose tolerance

Exclusion Criteria:

* HbA1c less than 6.5%
* Use of any glucose-lowering agents including metformin or sulfonylureas.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in beta-cell responsivity induced by glucagon | Beta-cell responsivity will be calculated as the gradient of the relationship between glucose concentrations and insulin secretion rate during the study day over the 4 hours (0 to 240 minutes) of the study
  The beta-cell responsivity observed during glucagon infusion will be compared to that observed during glucose infusion

SECONDARY OUTCOMES:
change in endogenous glucose production induced by glucagon | The rate of endogenous glucose production at the end of the study (240 minutes) will be expressed as a percentage of that at the beginning of the study (0 minutes). The % change for each study day will then be compared
  The endogenous glucose production observed during glucagon infusion will be compared to that observed during glucose infusion
change in glucose disappearance induced by glucagon | The rate of glucose disappearance at the end of the study (240 minutes) will be expressed as a percentage of that at the beginning of the study (0 minutes). The % change for each study day will then be compared
  The glucose disappearance observed during glucagon infusion will be compared to that observed during glucose infusion

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to the patient-level data, the metadata, data dictionary, statistical analysis plan, and final protocol will be shared. The sharing of the data dictionary, statistical analysis plan and final protocol with amendments will enable researchers to understand how the data was collected and to correctly interpret the data for future secondary analysis. We plan to share datasets resulting from the proposed studies in Vivli, a non-profit institution that supports the Vivli repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data shared will be archived and available on the platform for request by researchers for a minimum of 10 years after contribution. Data will be made accessible no later than the time of our associated publication or the end of the grant period (whichever comes first). On an ongoing basis, Vivli evaluates its data holdings regarding maintaining access and reserves the right to discontinue the distribution of a data collections when deemed appropriate. When materials are deaccessioned, the data are no longer publicly accessible at Vivli, they may still be preserved in Vivli's storage vault. Because digital files are assigned a persistent digital object identifier (DOI), the study description is still available to view, but is not searchable through Vivli.
Access Criteria: The data being shared is human data from clinical trials and therefore a higher level of protection is required. Access to this data will be controlled by a managed access process whereby access is provided only after approval. Data will be controlled access with the General Research Use Data Use Limitation, as allowed by the informed consent and the institutional certification.